CLINICAL TRIAL: NCT05558605
Title: Use of Artificial Intelligence-Guided Echocardiography to assIst cardiovascuLar Patient managEment
Acronym: AGILE-Echo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Collaborators: Alice Springs Hospital (Unknown); Princess Alexandra Hospital, Brisbane, Australia (Other); Royal Perth Hospital (Other); Ochre Health (Unknown); Walgett Aboriginal Medical Services (Unknown); Merriden Health Service (Unknown); Royal Hobart Hospital (Other Government); Quairading Medical Practice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 325-22
Record Dates: First submitted 2022-09-11; First posted 2022-09-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Valve Heart Disease
Keywords: Artificial intelligence; Echocardiography; Heart failure; Valve disease
MeSH Terms: conditions — Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Multicentre RCT comparing AI-TTE with usual care
Who Masked: Outcomes Assessor
Masking Description: PROBE design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Screening/Management Plan (Experimental): AI-guided echo acquisition performed using a desktop echo machine (uSmart 3300, Terason, Burlington, MA) with AI software (Caption Health, Brisbane, CA) obtained by a non-expert (eg. clinic nurse, registrar general practitioner or physician) at the remote clinic, usually on the day of clinic review. Images will then be uploaded onto a secure cloud and downloaded at the core lab for measurement, interpretation and reporting.
  Interventions: Diagnostic Test: AI-guided echo
- Usual care (Active Comparator): Standard echo acquisition by a sonographer either at a referral hospital, or by a visiting team - usually necessitating a delay. Measurement, interpretation and reporting will happen as usual.
  Interventions: Diagnostic Test: Standard echo

INTERVENTIONS:
Diagnostic Test: AI-guided echo — AI-guided echocardiography
  Arms: Screening/Management Plan
Diagnostic Test: Standard echo — Standard echocardiography
  Arms: Usual care

SUMMARY:
Heart Failure and valvular heart disease are disproportionate problems in rural and remote Australia (RRA). Echocardiography is the best imaging investigation, and essential for management, but access to this essential test shows huge geographic variations, primarily because of dependence on expert acquisition. This trial seeks to demonstrate the effectiveness of artificial intelligence-based echocardiography for triage and management of patients with known or suspected heart disease in RRA.

DETAILED DESCRIPTION:
Heart Failure (HF) and valvular heart disease (VHD) are disproportionate problems in rural and remote Australia (RRA) relative to the rest of the country, due in part to an ageing rural population and to the frequency of rheumatic heart disease in the Aboriginal community. Late diagnoses can lead to avoidable hospital admissions and expense to the Australian health system. Echocardiography is the imaging investigation of choice, and a cornerstone of management, but access to this essential test shows huge geographic variations in Australia. The primary reason for this is the dependence of this technique on expert acquisition. Artificial intelligence (AI) has now been harnessed to optimise echocardiographic image acquisition, and secure, cloud-based storage enables remote measurement and interpretation. This trial seeks to demonstrate the effectiveness of AI-based echocardiography-guided triage and management of patients with known or suspected heart disease in RRA. This study will involve the conduct of a world-first randomised controlled trial of AI-testing and early intervention to detect early stages of HF and VHD, select appropriate management, reduce admissions and preserve functional status and quality of life. The study will be conducted with partipants in RRA, aged 40 years and older with at least one HF risk factor and recruited through clinic and community outreach in four sites with the involvement of remote outreach from i) Alice Springs Hospitals, ii) Nepean Hospital to Dubbo Hospital and Western NSW, iii) Princess Alexandra Hospital to Roma, Charleville and Western Queensland, and iv) Perth Aboriginal communities in partnership with the Royal Perth hospital and the Derbarl Yerrigan Health Service. Approximately 1200 individuals at risk for HF and VHD will be screened and followed up. The study will be conducted in partnership with Aboriginal community partners.

ELIGIBILITY:
Inclusion Criteria:

* Age >45 years
* eligible for Medicare
* exercise intolerance or cardiovascular (CV) risk factors

Exclusion Criteria:

* Known HF or HVD
* situations where cardio-protection is already indicated (eg. known CAD)
* comorbid conditions with life expectancy <2 years
* inability to provide written informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of cardiac dysfunction or heart valve disease | 12 months
  Number of Participants with Diagnosis of cardiac dysfunction or heart valve disease

CONTACTS AND LOCATIONS:
Overall Officials: Tom Marwick, MBBS, PhD, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Alice Springs Hospital, Alice Springs, Northern Territory, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT05558605/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT05558605/ICF_001.pdf